CLINICAL TRIAL: NCT04700969
Title: Onset PrevenTIon of Urinary Retention in Orthopaedic Nursing and Rehabilitation, OPTION - a Knowledge Implementation Study on a Facilitation Strategy for Multi-professional Clinical Champion Teams
Brief Title: Onset PrevenTIon of Urinary Retention in Orthopaedic Nursing and Rehabilitation
Acronym: OPTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Linkoeping University (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ORU 2020/03330
Record Dates: First submitted 2020-12-23; First posted 2021-01-08 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Urinary Retention; Hip Fractures; Hip Arthritis
Keywords: Orthopedics; Implementation; Research utilization
MeSH Terms: conditions — Urinary Retention; Hip Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A support program to facilitate implementation of EBP for postoperative urinary retention (Experimental): 12- month support program. Multi-professional facilitator-teams will be supported by a 12-month support program including seminars and monthly supervision (e-discussion forum and group teleconferences) to develop an awareness of, and skills in facilitating implementation of evidence/EBP in clinical everyday care.
  Interventions: Other: : A support program to facilitate implementation of evidence-based practice for postoperative urinary retention
- Control-No support program (No Intervention): No support program

INTERVENTIONS:
Other: : A support program to facilitate implementation of evidence-based practice for postoperative urinary retention — A 12-month implementation support program for multi-professional internal facilitator teams
  Arms: A support program to facilitate implementation of EBP for postoperative urinary retention

SUMMARY:
Urinary retention (UR) is a common problem in older people undergoing hip surgery. Untreated UR can lead to bladder distention and a permanent damage of the bladder, which can cause both physical and psychical suffering as well as increased costs for society. Even if national and international practice guidelines are in place for handling UR within the health care system, many fail to comply with them. Compliance to clinical practice guidelines are improved if different professions and managers collaborate as a team. In OPTION (Onset PrevenTIon of urinary retention in Orthopedic Nursing and rehabilitation) the investigators will coach multi-professional local facilitator teams in knowledge translation and implementation of UR practice as well as investigate the effects of such evidence-based practice in orthopedic nursing and rehabilitation.

Implementation of research-based knowledge in evidence-based practice within an organization is complex with several known interacting factors. In a health care system these factors can be the care context, knowledge (innovation) and how the organization facilitates such implementations. The implementation strategy of OPTION utilize established theories of facilitation of knowledge implementation considering evidence and context with focus on leadership. The intervention consists of seminars and systematic support for implementation of UR-guidelines OPTION combine studies of adherence to evidence based practice regarding UR for patients over 65 years old that has undergone hip surgery and the health economic aspects of it. OPTION also contribute with improvements and increased knowledge regarding strategies to implement evidence based health care that can be used in other areas than UR and hip surgeries.

ELIGIBILITY:
Inclusion Criteria: Orthopaedic units in Sweden performing hip surgery. -

Exclusion Criteria: Orthopaedic units in Sweden not performing hip surgery

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to UR guidelines in the care of patients undergoing hip surgery. | Change from base line to 1 year after the intervention
  Adherence to national urinary retention guidelines documented in the patients' medical record

SECONDARY OUTCOMES:
Number of hip surgery patients with UR | Change from base line to 1 year after the intervention
  Number of hip surgery patients with UR documented in the patients' medical record
Patient participation | Change from base line to 1 year after the intervention
  The Patient Preferences for Patient Participation tool (The 4Ps)
Costs related to UR | Change from base line to 1 year after the intervention
  Costs for device and labour for bladder scanning and urinary catheterization
The IFs', staff's, and managers' experience of UR care | Change from base line to 1 year after the intervention
  Investigated with qualitative interviews
The IFs', staff's, and managers' experience of the facilitation program | 1 year after the intervention
  Investigated with qualitative interviews
The experience of people undergoing hip surgery, regarding UR, UR care. | Change from base line to 1 year after the intervention
  Investigated with qualitative interviews
The impact of a knowledge translation support program on the peoples' experience of the above | Change from base line to 1 year after the intervention
  Investigated with qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hälleberg Nyman, PHD, Principal Investigator — Örebro University, Sweden
Locations (17):
- Sweden (17):
  - Sjukhuset Arvika, Arvika
  - Danderyds sjukhus, Danderyd
  - Höglandssjukhuset Eksjö, Eksjö
  - Enköpings lasarett, Enköping
  - Mälarsjukhuset, Eskilstuna
  - Karolinska University Hospital, Huddinge, Huddinge
  - Capio Ortopediska huset, Johanneshov
  - Karlskoga Lasarett, Karlskoga
  - Capio Specialistvård Motala, Motala
  - Vrinnevisjukhuset, Norrköping
  - Norrtälje Sjukhus, Norrtälje
  - Nyköpings lasarett, Nyköping
  - Örebro University Hospital, Örebro
  - Södertälje sjukhus, Södertälje
  - Södersjukhuset, Stockholm
  - Sjukhuset Torsby, Torsby
  - Västmanlands sjukhus, Västerås

REFERENCES:
- [Derived] Winberg M, Fjordkvist E, Joelsson-Alm E, Carlfjord S, Nyman MH, Eldh AC. Contextual Factors Affecting Evidence-Based Practice in Orthopaedic Nursing and Rehabilitation: A Mixed Methods Study. J Adv Nurs. 2025 Jul 19. doi: 10.1111/jan.70098. Online ahead of print. PMID 40682329
- [Derived] Fjordkvist E, Halleberg Nyman M, Winberg M, Joelsson-Alm E, Eldh AC. First-line managers' experience of guideline implementation in orthopaedic nursing and rehabilitation: a qualitative study. BMC Health Serv Res. 2024 Jul 31;24(1):871. doi: 10.1186/s12913-024-11353-w. PMID 39085940
- [Derived] Eldh AC, Joelsson-Alm E, Wretenberg P, Halleberg-Nyman M. Onset PrevenTIon of urinary retention in Orthopaedic Nursing and rehabilitation, OPTION-a study protocol for a randomised trial by a multi-professional facilitator team and their first-line managers' implementation strategy. Implement Sci. 2021 Jun 26;16(1):65. doi: 10.1186/s13012-021-01135-x. PMID 34174917